CLINICAL TRIAL: NCT03153488
Title: Attention Deficit Hyperactivity Disorder (ADHD) Prediction of Treatment Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000547
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Methylphenidate; Amphetamine; Attention Deficit Hyperactivity Disorder; Treatment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Methylphenidate (Experimental): Adult subjects (ages 18-45) receiving a Methylphenidate derivative medication
  Interventions: Radiation: MRI
- Amphetamine (Experimental): Adult subjects (ages 18-45) receiving an Amphetamine derivative medication
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — All participants will perform one MRI session before initiation of treatment. The imaging session will last about an hour including the structural and functional MRI portions. The subjects lie on a padded scanner couch in a dimly illuminated room, and wear foam earplugs to attenuate scanner sounds.

SUMMARY:
This is a 6-month trial in adults to find out if certain neuromarkers can predict individual treatment response to stimulant medications for Attention Deficit Hyperactivity Disorder (ADHD). Males and females, ages 18-45, will complete an MRI scan at MIT prior to beginning medication for ADHD as determined by a treating clinician outside the context of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults ages 18-55
* A diagnosis of DSM-V ADHD based on clinical assessment supported by the ADHD module of a structured diagnostic interview
* Proficiency in English
* Right-handed

Exclusion Criteria:

* Any contraindication for the use of a stimulant medication
* Investigator and his/her immediate family (spouse, parent, child, grandparent, or grandchild)
* Any contraindications for MRI examination (metallic implants, such as pacemakers, surgical aneurysm clips, or known metal fragments in the body)
* Women who are currently pregnant or breastfeeding, as confirmed by a urine pregnancy test
* Clinically significant abnormal baseline laboratory values, including systolic and diastolic blood pressure parameters above 140 and 90, respectively and resting heart rate outside 60-100 bpm

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
ADHD Clinical Global Impressions Scale - Severity (CGI-S) | 6 months
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment.
ADHD Clinical Global Impressions Scale - Improvement (CGI-I) | 6 months
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.

SECONDARY OUTCOMES:
Connectomic Variation Prediction of Medicine Response | 6 months
  Examine whether variation in baseline ADHD severity scores and functional connectivity and structural connectivity predict whether an individual ADHD patient will respond better to one of the other stimulant family treatment, both, or neither. An MRI will be completed prior to starting medication.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States